CLINICAL TRIAL: NCT05089786
Title: Assessment of Safety and Feasibility of Exablate Neuro System to Perform Echo-Focusing Echo Imaging in Patients With Treatment-Resistant Neurologic and Psychiatric Indications
Brief Title: Echo-Focusing in Patients With Treatment-Resistant Neurologic and Psychiatric Indications (EF001)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: InSightec (Industry)
Collaborators: Health Canada (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EF001
Record Dates: First submitted 2021-09-22; First posted 2021-10-22 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Essential Tremor; Neurology
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-arm, non-randomized, feasibility trial with no control group seeks to evaluate the safety and efficacy of using the Exablate 4000 Type 1 or 1.1 System with Echo-focusing in patients with Major Depressive Disorder (MDD), Obsessive Compulsive Disorder (OCD), Essential Tremor (ET), Post Traumatic Stress Disorder (PTSD), anorexia nervosa (AN).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exablate Neuro System Treatment (Experimental): MR-Guided Focused Ultrasound with Echo-Focusing will be used to ablate a target area selected by the physician.
  Interventions: Device: Exablate Neuro Type 1.0 System with Echo Focusing

INTERVENTIONS:
Device: Exablate Neuro Type 1.0 System with Echo Focusing — MR-Guided Focused Ultrasound
  Other Names: Focused Ultrasound; MRgFUS; FUS

SUMMARY:
Evaluate the safety and effectiveness of Echo-Focusing using Exablate Neuro as a tool for treating patients with treatment-refractory neurologic and psychiatric disorders.

DETAILED DESCRIPTION:
The objective of the proposed study is to evaluate the safety and effectiveness of Echo-Focusing using Exablate Neuro as a tool for treating patients with treatment-refractory neurologic and psychiatric disorders. Safety will be determined by an evaluation of the incidence and severity of procedure-related complications from the treatment day visit through the 12-month post-treatment time point, although events that are not procedure or device related will be also captured and recorded. Clinical efficacy will be determined using standard clinical metrics, appropriate for the patient's condition.

The hypotheses tested include:

1. Exablate ablation with Echo-Focusing can be safely performed in patients suffering from treatment-resistant psychiatric illness and essential tremor.
2. Echo-Focusing will allow for more efficient (faster) treatments, which require less energy (measured in Joules), as compared to published data from Exablate thalamotomy99 and Exablate-capsulotomy100 performed without Echo-Focusing.
3. Lesion appearances following Exablate ablation with Echo-Focusing will be similar in radiographic appearance to those created without Echo-Focusing.
4. Patients who undergo Exablate ablation with Echo-Focusing will demonstrate similar rates of clinical improvement from those seen after non-Echo-Focusing ablation.

ELIGIBILITY:
Inclusion Criteria: - Inclusion Criteria for Major Depressive Disorder (MDD):

1. Men and women ≥ 20 and ≤ 80 years of age.
2. Patients who are able and willing to give consent and physically and practically able to attend study visits, as determined by both study psychiatrist and the surgeon.
3. DSM-V diagnosis of major depressive disorder (MDD), or bipolar disorder with predominant depressive symptoms.
4. At least 5-year illness history of the primary disorder and at least 6 months since the onset of the first episode of major depression.
5. A minimum score of 20 on the Hamilton Depression Rating Scale (HAMD) when depressed (patients with bipolar disorder may be rapid cycling, but must have at least 2 weeks of major depression at the time the HAMD is conducted).
6. Medication-refractoriness as determined by an adequate dose and duration of standard psychiatric treatments (including psychotherapy and/or pharmacology) as determined by a psychiatrist associated with the study. Including specifically:

   1. Failed to respond or tolerate adequate trials of three or more medications accepted as first line therapies in the treatment of depression.
   2. Failed to respond or tolerate augmentation with or combination of at least 2 medications known to be first line treatments for depression.
   3. An adequate trial of Cognitive Behavioural Therapy (CBT) or other evidence-supported psychotherapy, delivered by a therapist experienced in treating depression.
7. Able to communicate sensations during the Exablate MRgFUS treatment.
8. A consistent dose of any and all medications in the 30 days prior to study entry.
9. Women of childbearing potential must agree to use a contraception method throughout the study.

Inclusion Criteria for Obsessive Compulsive Disorder (OCD):

1. Men and women ≥20 and ≤80 years of age.
2. Patients who are able and willing to give consent and physically and practically able to attend study visits, as determined by both study psychiatrist and the surgeon.
3. DSM-V diagnosis of Obsessive-Compulsive Disorder (OCD), at least 5-year illness history with a minimum score of 28 on the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS).
4. Medication-refractoriness as determined by an adequate dose and duration of standard psychiatric treatments (including psychotherapy and/or pharmacology) as determined by a psychiatrist associated with the study. Including specifically:

   1. Failed adequate trial of three or more medications accepted as first line therapies in the treatment of OCD.
   2. Attempted augmentation, if tolerated, by at least 2 medications known to be first line treatments for OCD.
5. An adequate trial of CBT, delivered by a therapist experienced in treating OCD.
6. A consistent dose of all medications in the 30 days prior to study entry.
7. Able to communicate sensations during the Exablate MRgFUS treatment.
8. Women of childbearing potential must agree to use a contraception method throughout the study.

Inclusion Criteria for Post Traumatic Stress Disorder (PTSD):

1. Men and women ≥ 20 and ≤ 80 years of age.
2. Patients who are able and willing to give consent and physically and practically able to attend study visits, as determined by both study psychiatrist and the surgeon.
3. Diagnosis of Post-Traumatic Stress Disorder and Major Depressive Disorder, as defined by the Diagnostic and Statistical Manual fifth edition (DSM V).
4. Severe PTSD symptoms, as measured by Clinician Administered PTSD scale (CAPS) scores ≥ 50.
5. Treatment Resistance as defined by the persistence of clinical symptoms despite adequate treatment with four modalities, including a) selective serotonin reuptake inhibitors, b) cognitive behavioral therapy, c) other classes of medications and/or psychotherapy.
6. DSM-V diagnosis of major depressive disorder with at least 5 years illness history .
7. A minimum score of 20 on the Hamilton Depression Rating Scale (HAMD).
8. A pattern of chronic stable PTSD lasting at least 1 year.
9. Able to communicate sensations during the Exablate MRgFUS treatment.
10. A consistent dose of any and all medications in the 30 days prior to study entry.
11. Women of childbearing potential must agree to use a contraception method throughout the study.

Inclusion Criteria for Anorexia Nervosa (AN):

1. Men and women ≥ 20 and ≤ 80 years of age.
2. Patients who are able and willing to give consent and physically and practically able to attend study visits, as determined by both study psychiatrist and the surgeon.
3. DSM-V diagnosis of anorexia nervosa, restricting or binge-purging subtype.
4. Chronicity of treatment resistance shown by some or all of:

   1. A pattern of 3 years' duration of relentless unresponsiveness to ≥ 2 voluntary hospital admissions, characterized by failure to complete treatment or immediate weight relapse after treatment
   2. A pattern of increasing medical instability, accompanied by refusal to participate in or a pattern of poor response to intensive expert treatment and increasing medical acuity, lasting at least 2 years, and including at least 2 episodes of involuntary feeding.
   3. A pattern of chronic stable anorexia nervosa that has lasted at least 10 years.
5. DSM-V diagnosis of major depressive disorder OR obsessive-compulsive disorder with at least 5 years illness history:

   a. If MDD diagnosis, HAMD > 20; if OCD diagnosis, YBOCS ≥ 28.
6. Treatment refractory to either MDD or OCD, with documented non-response to three primary medication trials, 2 augmentation trials, and at least one completed course of CBT.
7. Potassium levels within normal laboratory range.
8. Able to communicate sensations during the Exablate MRgFUS treatment.
9. A consistent dose of any and all medications in the 30 days prior to study entry.
10. Women of childbearing potential must agree to use a contraception method throughout the study.

Inclusion Criteria for Essential Tremor:

1. Men and women ≥ 20 and ≤ 80 years of age.
2. Patients who are able and willing to give consent and physically and practically able to attend study visits, as determined by both study neurologist and the surgeon.
3. A confirmed diagnosis of Essential Tremor by a neurologist.
4. Refractory to at least two trials of medication therapy, including at least one first-line agent (propranolol or primidone).
5. Able to communicate sensations during the Exablate MRgFUS treatment.
6. A consistent dose of any and all medications in the 30 days prior to study entry.
7. Women of childbearing potential must agree to use a contraception method throughout the study.

Exclusion Criteria (Common for all Cohorts):

1. Patients with unstable cardiac status [e.g., unstable angina pectoris on medication, patients with documented myocardial infarction within six months, congestive heart failure requiring medication (other than diuretics), patients on anti-arrhythmic drugs, severe hypertension (defined as systolic blood pressure > 150 mm Hg or diastolic blood pressure > 100 mm Hg while on medication)].
2. Patients with standard contraindications for MRI imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
3. Severely impaired renal function (estimated glomerular filtration rate < 30 ml/min/1.73 m2) or receiving dialysis.
4. Laboratory biochemical evidence of abnormal bleeding and/or coagulopathy, including risk factors for intraoperative or postoperative bleeding (platelet count less than 100,000 per cubic millimeter or abnormal INR).
5. Cerebrovascular disease (e.g., CVA within 6 months) or history of intracranial hemorrhage.
6. Untreated, uncontrolled sleep apnea.
7. Receiving anticoagulant (e.g., warfarin) or antiplatelet (e.g., aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g., Avastin) within one month of focused ultrasound procedure.
8. Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment.
9. Patients unable to communicate with the investigator and staff.
10. Presence of significant cognitive impairment.
11. Presence of psychosis on clinical evaluation.
12. Patients with brain tumors already known or revealed on pretreatment MRI.
13. Currently pregnant (as determined by history and serum HCG) or lactating.
14. Patients who have right-to-left, bidirectional, or transient right-to-left cardiac shunts.
15. Patients with relative contraindications to DEFINITY ultrasound contrast agent including subjects with a family or personal history of QT prolongation or taking concomitant medications known to cause QTc prolongation (QT prolongation observed on screening ECG (QTc > 450 for men and >470 for women).
16. Currently admitted as an inpatient to a medical facility.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-12-31 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events | Time of Exablate transcranial procedure
  Safety will be assessed by evaluating the incidence and severity of device and procedure related adverse events
Change in Quality of Life per the Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (QLESQ-SF) | 12 months
  Clinical efficacy will be assessed by evaluating change in quality of life per the Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (QLESQ-SF). This 16-item self-report rating inventory measures the degree of enjoyment and satisfaction experienced by subjects in various areas of daily functioning (scale 1 to 5). A higher total score correlates with greater satisfaction. The survey will be collected before and after treatment at day 1 and months 1, 3, 6, and 12 to determine any effect and its change over time.